CLINICAL TRIAL: NCT04672954
Title: Pharmacokinetics and Pharmacodynamic Effects of Different Single Oral Doses of BI 474121 in Healthy Male Subjects
Brief Title: A Study in Healthy Men to Test How Different Doses of BI 474121 Are Taken up and How They Influence the Amount of a Molecular Messenger (cGMP) in the Spinal Fluid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1411-0013; 2020-002321-28 (EudraCT Number)
Record Dates: First submitted 2020-12-14; First posted 2020-12-17 (Actual); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-07

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: This trial is designed to have three parts. Part 1: single-blind, randomized, placebo-controlled. Part 2: open-label, non-randomized. Part 3: open-label, randomized.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo matching to 10 mg BI 474121 administered as uncoated tablets with 240 milliliter of water after subjects fasted overnight for at least 10 hours. This arm was part of Part 1: randomised, placebo-controlled, single-blind.
  Interventions: Drug: Placebo
- 2.5 milligram (mg) BI 474121 (Experimental): 2.5 mg BI 474121 administered as uncoated tablets (1 x 2.5 mg) with 240 milliliter of water after subjects fasted overnight for at least 10 hours. This arm was part of Part 3 of the study: randomised, open-label.
  Interventions: Drug: 2.5 milligram (mg) BI 474121
- 10 milligram (mg) BI 474121 (Experimental): 10 mg BI 474121 administered as uncoated tablets (1 x 10 mg) with 240 milliliter of water after subjects fasted overnight for at least 10 hours. This arm was part of Part 3 of the study: randomised, open-label.
  Interventions: Drug: 10 milligram (mg) BI 474121
- 20 milligram (mg) BI 474121 (Experimental): 20 mg BI 474121 administered as uncoated tablets (2 x 10 mg) with 240 milliliter of water after subjects fasted overnight for at least 10 hours. This arm was part of Part 1 of the study: randomised, placebo-controlled, single-blind.
  Interventions: Drug: 20 milligram (mg) BI 474121
- 40 milligram (mg) BI 474121 (Experimental): 40 mg BI 474121 administered as uncoated tablets (4 x 10 mg) with 240 milliliter of water after subjects fasted overnight for at least 10 hours. This arm was part of Part 2 of the study: non-randomised, open-label.
  Interventions: Drug: 40 milligram (mg) BI 474121

INTERVENTIONS:
Drug: Placebo — Placebo matching to 10 mg BI 474121 administered as uncoated tablets with 240 milliliter of water after subjects fasted overnight for at least 10 hours. This arm was part of Part 1: randomised, placebo-controlled, single-blind.
  Arms: Placebo
Drug: 2.5 milligram (mg) BI 474121 — 2.5 mg BI 474121 administered as uncoated tablets (1 x 2.5 mg) with 240 milliliter of water after subjects fasted overnight for at least 10 hours. This arm was part of Part 3 of the study: randomised, open-label.
  Arms: 2.5 milligram (mg) BI 474121
Drug: 10 milligram (mg) BI 474121 — 10 mg BI 474121 administered as uncoated tablets (1 x 10 mg) with 240 milliliter of water after subjects fasted overnight for at least 10 hours. This arm was part of Part 3 of the study: randomised, open-label.
  Arms: 10 milligram (mg) BI 474121
Drug: 20 milligram (mg) BI 474121 — 20 mg BI 474121 administered as uncoated tablets (2 x 10 mg) with 240 milliliter of water after subjects fasted overnight for at least 10 hours. This arm was part of Part 1 of the study: randomised, placebo-controlled, single-blind.
  Arms: 20 milligram (mg) BI 474121
Drug: 40 milligram (mg) BI 474121 — 40 mg BI 474121 administered as uncoated tablets (4 x 10 mg) with 240 milliliter of water after subjects fasted overnight for at least 10 hours. This arm was part of Part 2 of the study: non-randomised, open-label.
  Arms: 40 milligram (mg) BI 474121

SUMMARY:
The main objectives of this trial are:

* To evaluate the effect of BI 474121 on cyclic guanosine monophosphate (cGMP) levels in cerebrospinal fluid (CSF)
* To assess the exposure of BI 474121 in CSF relative to plasma
* To determine the exposure effect relationship in CSF with different oral doses of BI 474121

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 65 years (inclusive)
* BMI of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 150 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders assessed as clinically relevant by the investigator
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Further exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] van Kraaij S, Goeldner RG, Rosenbrock H, Groeneveld GJ, Kremer P, Schaible J, Zambori J, Schultheis C. Effects of the phosphodiesterase 2 inhibitor BI 474121 on central nervous system cyclic guanosine monophosphate concentrations: Translational studies. Br J Clin Pharmacol. 2024 Oct;90(10):2517-2528. doi: 10.1111/bcp.16137. Epub 2024 Jun 16. PMID 38880932
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of three parts, part 1: randomised, placebo-controlled, single-blind, part 2:non-randomised, open-label and part 3: randomised, open-label, with the aim of exploring the pharmacokinetics and pharmacodynamic effects of different single oral doses of BI 474121 in healthy male subjects
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Placebo | 2.5 Milligram (mg) BI 474121 | 10 Milligram (mg) BI 474121 | 20 Milligram (mg) BI 474121 | 40 Milligram (mg) BI 474121
Started | 4 | 4 | 4 | 6 | 6
Completed | 4 | 4 | 4 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): all subjects who were entered and treated with one dose of study drug (i.e. verum or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 2.5 Milligram (mg) BI 474121 | 10 Milligram (mg) BI 474121 | 20 Milligram (mg) BI 474121 | 40 Milligram (mg) BI 474121 | Total
Number analyzed (Participants) | 4 | 4 | 4 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (24.3) | 27.5 (9.3) | 22.0 (3.2) | 38.3 (17.4) | 23.2 (2.9) | 30.5 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 4 | 4 | 4 | 6 | 6 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 4 | 3 | 4 | 6 | 6 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 1
  White | 4 | 3 | 4 | 5 | 5 | 21
  More than one race | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Exposure-related Change From Baseline (Calculated as Ratio) of Cyclic Guanosine Monophosphate (cGMP) in Cerebrospinal Fluid (CSF)
Description: Maximum exposure-related change from baseline (calculated as ratio) of cyclic guanosine monophosphate (cGMP) in Cerebrospinal fluid (CSF). In subjects treated with BI 474121 this is the maximum cGMP value measured within 1 hour (h) prior and 4 h post BI 474121 Maximum measured concentration (Cmax) in CSF. For subjects treated with placebo, this is the maximum cGMP value measured within 1 h prior to and 4 h after the median BI 474121 tmax (time from (last) dosing to the maximum measured concentration of the analyte) in CSF of the BI 474121 treated subjects. Baseline cGMP concentration was calculated as the arithmetic mean of all pre-dose measurements above Lower limit of quantification (LLOQ) obtained in that subject. The maximum exposure-related change from baseline in cGMP in CSF was explored using an analysis of covariance (ANCOVA) model on the logarithmic scale. Maximum exposure related cGMP: Ratio [maximum cGMP / baseline cGMP].
Time Frame: Within approximately 2, 1, and 0.17 hours before and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14 and 24 hours following drug administration.
Population: Pharmacodynamic parameter analysis set (PDS): all evaluable subjects who were entered and treated with one dose of study drug and who provided at least one evaluable pre- and post-dose measure for a pharmacodynamic endpoint.
Measure: Geometric Mean (Standard Error); unit: maximum change from baseline cGMP ratio
Arm/Group | Placebo | 2.5 Milligram (mg) BI 474121 | 10 Milligram (mg) BI 474121 | 20 Milligram (mg) BI 474121 | 40 Milligram (mg) BI 474121
Number analyzed (Participants) | 4 | 4 | 4 | 6 | 5
maximum change from baseline cGMP ratio | NA (NA) — Geometric Mean is adjusted Geometric Mean = 1.26 Standard Error is Geometric standard error (gSE) = 1.24 | NA (NA) — Geometric Mean is adjusted Geometric Mean = 1.62 Standard Error is Geometric standard error (gSE) = 1.23 | NA (NA) — Geometric Mean is adjusted Geometric Mean = 2.09 Standard Error is Geometric standard error (gSE) = 1.23 | NA (NA) — Geometric Mean is adjusted Geometric Mean = 1.44 Standard Error is Geometric standard error (gSE) = 1.18 | NA (NA) — Geometric Mean is adjusted Geometric Mean = 2.20 Standard Error is Geometric standard error (gSE) = 1.20
Statistical Analysis 1: Comparison: Placebo vs 2.5 Milligram (mg) BI 474121; The difference between the expected means for ln(T) - ln(R) was estimated by the difference in the corresponding least square means (point estimate) and two-sided 90% confidence intervals based on the t-distribution were computed. These quantities were back-transformed to the original scale to give the point estimator and interval estimates; Test type: Other; p = 0.3941, ANCOVA; Ratio = 1.29, 90% CI 2-sided [0.78 to 2.13] — Ratio = BI / Placebo. Geometric standard error = 1.34
Statistical Analysis 2: Comparison: Placebo vs 10 Milligram (mg) BI 474121; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.1089, ANCOVA; Ratio = 1.66, 90% CI 2-sided [0.99 to 2.79] — Ratio = BI / Placebo. Geometric standard error = 1.35
Statistical Analysis 3: Comparison: Placebo vs 20 Milligram (mg) BI 474121; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.6308, ANCOVA; Ratio = 1.14, 90% CI 2-sided [0.71 to 1.85] — Ratio = BI / Placebo. Geometric standard error = 1.32
Statistical Analysis 4: Comparison: Placebo vs 40 Milligram (mg) BI 474121; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0690, ANCOVA; Ratio = 1.75, 90% CI 2-sided [1.06 to 2.89] — Ratio = BI / Placebo. Geometric standard error = 1.33

2. Primary Outcome: Maximum Measured Concentration (Cmax) Ratio of BI 474121 in Cerebrospinal Fluid (CSF) Compared to Plasma
Description: Maximum measured concentration (Cmax) ratio of BI 474121 in CSF compared to plasma. Mixed effects model: random effect 'subject nested within treatment', fixed effect, treatment, substance and their interaction' (for estimation of overall group effect the model was run without interaction term). Cmax was log transformed (natural logarithm) prior to fitting the model. Difference between expected means for log(CSF)- log(plasma) was estimated by difference in the corresponding least square means (point estimate) and two-sided 90% CI based on the t-distribution were computed. Quantities were back-transformed to the original scale to give an point estimator and interval estimate. Ratio = CSF (T) / plasma (R).
  Plasma: Within 3 hours (h) before and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24, 34, 48 and 72 h following drug administration.
  CSF: Within approximately 2, 1, and 0.17 h before and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14 and 24 h following drug administration.
Time Frame: Up to 72 hours, see endpoint description for detailed sampling scheme.
Population: Pharmacokinetic parameter analysis set (PKS): This set includes all subjects who were entered and treated with one dose of study drug and who provide at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio [%] Cmax CSF (T) / Cmax Plasma (R)
Groups:
- Overall BI 474121: All dose groups of BI 474121 administered as uncoated tablets with 240 milliliter of water after subjects fasted overnight for at least 10 hours.
Arm/Group | 2.5 Milligram (mg) BI 474121 | 10 Milligram (mg) BI 474121 | 20 Milligram (mg) BI 474121 | 40 Milligram (mg) BI 474121 | Overall BI 474121
Number analyzed (Participants) | 4 | 4 | 6 | 5 | 19
Ratio [%] Cmax CSF (T) / Cmax Plasma (R) | 9.49 [8.27 to 10.89] | 7.88 [6.86 to 9.04] | 9.89 [8.84 to 11.07] | 8.42 [7.45 to 9.53] | 8.96 [8.37 to 9.59]

3. Secondary Outcome: Maximum Measured Concentration (Cmax) of BI 474121 in Plasma
Description: Maximum measured concentration (Cmax) of BI 474121 in plasma.
Time Frame: Within 3 hours before and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24, 34, 48 and 72 hours following drug administration.
Population: Pharmacokinetic parameter analysis set (PKS): This set includes all subjects who were entered and treated with one dose of study drug and who provide at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject will be included in the PKS, even if he/she contributes only one PK parameter value to the statistical assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomol/Liter
Arm/Group | 2.5 Milligram (mg) BI 474121 | 10 Milligram (mg) BI 474121 | 20 Milligram (mg) BI 474121 | 40 Milligram (mg) BI 474121
Number analyzed (Participants) | 4 | 4 | 6 | 5
Nanomol/Liter | 22.0 (30.0) | 87.2 (30.3) | 137 (21.7) | 278 (13.4)

4. Secondary Outcome: Maximum Measured Concentration (Cmax) of BI 474121 in Cerebrospinal Fluid (CSF)
Description: Maximum measured concentration (Cmax) of BI 474121 in Cerebrospinal fluid (CSF).
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomol/Liter
Arm/Group | 2.5 Milligram (mg) BI 474121 | 10 Milligram (mg) BI 474121 | 20 Milligram (mg) BI 474121 | 40 Milligram (mg) BI 474121
Number analyzed (Participants) | 4 | 4 | 6 | 5
Nanomol/Liter | 2.09 (27.9) | 6.87 (25.9) | 13.6 (9.17) | 23.5 (25.0)

5. Secondary Outcome: Time From Dosing to Maximum Measured BI 474121 Concentrations in Plasma (Tmax)
Description: Time from dosing to maximum measured BI 474121 concentrations in plasma (tmax).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | 2.5 Milligram (mg) BI 474121 | 10 Milligram (mg) BI 474121 | 20 Milligram (mg) BI 474121 | 40 Milligram (mg) BI 474121
Number analyzed (Participants) | 4 | 4 | 6 | 5
hours | 4.00 [1.50 to 5.02] | 1.50 [1.00 to 3.00] | 2.01 [1.00 to 3.00] | 4.00 [1.50 to 5.08]

6. Secondary Outcome: Time From Dosing to Maximum Measured BI 474121 Concentrations in CSF (Tmax)
Description: Time from dosing to maximum measured BI 474121 concentrations in CSF (tmax).
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | 2.5 Milligram (mg) BI 474121 | 10 Milligram (mg) BI 474121 | 20 Milligram (mg) BI 474121 | 40 Milligram (mg) BI 474121
Number analyzed (Participants) | 4 | 4 | 6 | 5
hours | 2.03 [2.03 to 4.02] | 2.03 [1.02 to 3.02] | 3.02 [2.03 to 3.07] | 4.03 [2.03 to 5.12]

7. Secondary Outcome: Maximum Measured Exposure-related cGMP Concentration in Cerebrospinal Fluid (CSF)
Description: Maximum measured exposure-related cGMP concentration in CSF. In subjects treated with BI 474121 this is the maximum cGMP value measured within 1 hour (h) prior and 4 h post BI 474121 Maximum measured concentration (Cmax) in CSF. For subjects treated with placebo, this is the maximum cGMP value measured within 1 h prior to and 4 h after the median BI 474121 tmax (time from (last) dosing to the maximum measured concentration of the analyte) in CSF of the BI 474121 treated subjects.
Time Frame: as for outcome 1
Population: Pharmacodynamic parameter analysis set (PDS): This set includes all evaluable subjects who provide at least one evaluable pre- and post-dose measure for a PD endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomol/Liter
Arm/Group | Placebo | 2.5 Milligram (mg) BI 474121 | 10 Milligram (mg) BI 474121 | 20 Milligram (mg) BI 474121 | 40 Milligram (mg) BI 474121
Number analyzed (Participants) | 4 | 4 | 4 | 6 | 5
Nanomol/Liter | 7.51 (40.0) | 9.54 (32.5) | 10.7 (79.2) | 7.36 (40.4) | 11.1 (37.8)

ADVERSE EVENTS:
Time Frame: Adverse events: day of drug administration + 7 days, up to 7 days. All-cause mortality: day of drug administration till trial completion date, up to 14 days.
Description: Treated set (TS): The treated set includes all entered subjects who were treated with one dose of study drug (i.e. verum or placebo).
Arm/Group | Placebo | 2.5 Milligram (mg) BI 474121 | 10 Milligram (mg) BI 474121 | 20 Milligram (mg) BI 474121 | 40 Milligram (mg) BI 474121
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 4/4 | 6/6 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4) | 2.5 Milligram (mg) BI 474121 (N=4) | 10 Milligram (mg) BI 474121 (N=4) | 20 Milligram (mg) BI 474121 (N=6) | 40 Milligram (mg) BI 474121 (N=6)
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 4
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 1
Catheter site pain (General disorders) | 0 | 1 | 1 | 0 | 2
Fatigue (General disorders) | 0 | 1 | 2 | 0 | 0
Feeling hot (General disorders) | 0 | 1 | 1 | 0 | 0
Hangover (General disorders) | 0 | 0 | 1 | 0 | 0
Puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 3 | 4 | 4 | 5 | 5
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 2 | 2
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 0 | 2 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 1 | 0 | 2
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT04672954/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT04672954/SAP_001.pdf